CLINICAL TRIAL: NCT07243223
Title: Epidemiological Profiles, Traditional Chinese Medicine Syndrome, and Biomarkers of Urinary Incontinence in Older Hong Kong Women: A Cross-sectional Study
Brief Title: Urinary Incontinence in Older Hong Kong Women: A Cross-sectional Study
Acronym: PROMOTE
Status: Not yet recruiting | Type: Observational
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Prof., Hong Kong Baptist University
Other Study IDs: REC/24-25/0631
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Urinary Incontinence in Old Age
Keywords: urinary incontinence; female
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine, blood, and stool samples will be collected. Urine: urinalysis, urinary microbiome (16S sequencing), and metabolomics. Blood: routine tests, metabolic and inflammatory markers, transcriptomics (whole blood), metabolomics and proteomics (serum). Stool: routine tests, metabolomics, gut microbiome (16S sequencing). Analyses will explore associations between biospecimen profiles and urinary incontinence clinical features.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stress Urinary Incontinence (SUI): Women diagnosed with SUI per EAU and ICS criteria: involuntary leakage during increased intra-abdominal pressure (e.g., exertion, coughing), stopping when the activity ends. Confirmed by positive cough stress or 1-hour pad test (>1g leakage), and bladder diary showing stress-only leakage. Initial screening uses the Chinese 3IQ, option A ("leakage with physical activity"). Cases with urge or mixed symptoms are excluded. No intervention to be administered.
- Urge Urinary Incontinence (UUI): Women diagnosed with UUI per EAU and ICS criteria: involuntary leakage of urine accompanied by or immediately preceded by urgency. Preliminary screening with Chinese 3IQ, option B ("leakage with urgency"). Final diagnosis confirmed by a bladder diary showing urgency-only leakage. Cases with stress or mixed symptoms are excluded. No intervention to be administered.
- Mixed Urinary Incontinence (MUI): Women diagnosed with MUI per EAU and ICS guidelines: symptoms of both stress and urge urinary incontinence. Confirmed by positive 1-hour pad test (>1g) and bladder diary showing both stress- and urgency-related leakage. Preliminary screening with Chinese 3IQ, option D ("leakage equally with activity and urgency"). Cases with pure stress or urge incontinence excluded. No intervention to be administered.
- Healthy Volunteers (HC): Female volunteers aged ≥55, living in Hong Kong ≥1 year, no history or symptoms of urinary incontinence, no recent urological consultation, and no major comorbidities (except well-controlled hypertension/hyperlipidemia). Not using drugs affecting urination or the gut microbiota. Able to understand instructions and provide consent. Exclusions: UI diagnosis, involuntary urine leakage, severe illness interfering with assessment. No intervention to be administered.

SUMMARY:
This is a prospective, cross-sectional study aim to include 1000 patients with urinary incontinence and 100 healthy controls in Hong Kong. The overall objection is to address the gaps in epidemiological profiles, TCM syndrome differentiation, and biomarkers discovery of urinary incontinence among older women. The specific aims including:

1. To assess the epidemiological characteristics of urinary incontinence among older women, as well as patients' knowledge and healthcare-seeking barriers, and to explore factors influencing the disease subtypes, severity, and healthcare-seeking behaviors;
2. To establish diagnostic criteria for traditional Chinese medicine (TCM) syndrome differentiation of urinary incontinence, and analyze the distribution of TCM syndromes;
3. To explore diagnostic biomarkers and severity evaluation biomarkers for three subtypes of urinary incontinence (SUI, UUI, MUI).

DETAILED DESCRIPTION:
This study is a cross-sectional observational study designed in accordance with the STROBE (Strengthening the Reporting of Observational Studies in Epidemiology) guidelines. A total of 1,000 female patients with urinary incontinence and 100 healthy controls will be enrolled.

Both urinary incontinence group and healthy group will be recruited through a combination of online publicity (via social media platforms) and offline community outreach. Each participant will be scheduled for a visit, during which the research staff will introduce the study's objectives, procedures, nature, and data privacy policy. Informed consent will be obtained. Socio-epi-demographic information (including age, educational level, marital status, occupation, income, reproductive history, medical history, comorbidities, medication history, diagnosis and treatment for urinary incontinence) and the type, frequency and severity of lower urinary tract symptoms will be collected.

Then, eligible participants with symptoms of urinary incontinence will undergo a 1-hour pad test, bladder capacity and post-void residual volume measurements, and a 1-week bladder diary to confirm the subtype of urinary incontinence (SUI, MUI, UUI) and its severity (mild, moderate, severe). Standardized questionnaires will be administered to assess the cognitive level regarding urinary incontinence (UIQ), quality of life (IIQ-7 and ICIQ-UI-SF), and barriers to care seeking (Barriers to Incontinence Care Seeking Questionnaire). Hand grip strength test will be conducted to evaluate the muscle strength. The first 300 urinary incontinence patients (100 with SUI, 100 with UUI, and 100 with MUI) enrolled in the study, who do not have chronic comorbidities (except for well-controlled hypertension or hyperlipidemia) and are not taking medications that affect urination or gut microbiota, will proceed to TCM syndrome differentiation and bio-sample collection. TCM syndrome differentiation related symptoms and signs will be collected for Delphi consensus research and cluster analysis. Blood, urine, stool routine lab tests (including metabolic and inflammatory markers such as fasting blood glucose, fasting triglycerides, albumin, creatinine, glucose, C-reactive protein, white blood cell count, etc.) and biological sample collection will also be performed for these patients.

Eligible participants who have never experienced symptoms of urinary incontinence and have no chronic comorbidity (expect for well-controlled hypertension and hyperlipidemia) and are not taking medications that affect urination or gut microbiota will serve as healthy controls. For healthy group, only blood, urine, stool routine lab tests and bio-sample will be conducted.

All data will be independently collected and cross-verified by two researchers, and entered into the electronic data management system (REDCap).

ELIGIBILITY:
Diagnostic Criteria:

1. Urinary Incontinence (UI)：Urinary incontinence will be diagnosed according to the definition of the International Continence Society (ICS), that is, 'any involuntary leakage of urine'. In addition, participants must have experienced this symptom continuously for at least six months to exclude cases of transient urinary incontinence.

2. Stress Urinary Incontinence (SUI)：The clinical diagnosis of SUI will be made with reference to the guidelines of the European Association of Urology (EAU) and the International Continence Society (ICS):

1. Symptoms: Involuntary leakage of urine during activities that increase intra-abdominal pressure, such as physical exertion, laughing, coughing, or walking; urine leakage stops immediately when the activity ceases.
2. Signs: Positive result on the cough stress test or a positive 1-hour pad test (the procedure will follow the standardized ICS protocol; leakage >1g is considered positive).
3. Pure urge incontinence and mixed urinary incontinence will be excluded. This subtype will be preliminarily identified using the Chinese version of the "3 Incontinence Questions" (3IQ): "During the past three months, in which of the following situations did you most often experience urine leakage? (single choice) A. During physical activities such as coughing, sneezing, lifting, or exercise; B. When you had the urge to urinate or felt the need to empty your bladder but could not reach the toilet in time; C. Without physical activity or urge; D. Equally during physical activity and urgency." (Selection of option A) SUI will be finally confirmed by a one-week bladder diary (showing only stress-related leakage) and a positive 1-hour pad test.

3. Urge Urinary Incontinence (UUI)：The clinical diagnosis of UUI will follow the guidelines of the European Association of Urology (EAU) and the International Continence Society (ICS):

1. Symptoms: Involuntary leakage of urine accompanied by or immediately preceded by urgency (a sudden, compelling desire to void that is difficult to defer).
2. Cases of pure stress urinary incontinence and mixed urinary incontinence will be excluded.

This subtype will be preliminarily identified using the Chinese version of the "3 Incontinence Questions" (3IQ): "During the past three months, in which of the following situations did you most often experience urine leakage? (single choice) A. During physical activities such as coughing, sneezing, lifting, or exercise; B. When you had the urge to urinate or felt the need to empty your bladder but could not reach the toilet in time; C. Without physical activity or urge; D. Equally during physical activity and urgency." (Selection of option B) Final confirmation will be based on a one-week bladder diary recorded by the participant (showing only urgency-related leakage).

4. Mixed Urinary Incontinence (MUI)：The clinical diagnosis of MUI will follow the guidelines of the European Association of Urology (EAU) and the International Continence Society (ICS):

1. Symptoms: The presence of stress urinary incontinence symptoms, such as involuntary leakage of urine during activities that increase intra-abdominal pressure (e.g., exercise, laughing, coughing, walking), with urine flow ceasing immediately upon stopping the activity; and, at the same time, the presence of urge urinary incontinence symptoms, such as urgency (a sudden, compelling desire to void that is difficult to defer) accompanied by or immediately followed by involuntary leakage of urine.
2. Signs: Positive result on the cough stress test or a positive 1-hour pad test (the procedure will follow the standardized protocol of the ICS; leakage >1g is considered positive).
3. Cases of pure urge urinary incontinence and pure stress urinary incontinence will be excluded.

This subtype will be preliminarily identified using the Chinese version of the "3 Incontinence Questions" (3IQ): "During the past three months, in which of the following situations did you most often experience urine leakage? (single choice) A. During physical activities such as coughing, sneezing, lifting, or exercise; B. When you had the urge to urinate or felt the need to empty your bladder but could not reach the toilet in time; C. Without physical activity or urge; D. Equally during physical activity and urgency." (Selection of option D) Final confirmation will be based on a one-week bladder diary recorded by the participant (showing both urgency- and stress-related leakage) and a positive 1-hour pad test.

5. Inclusion Criteria for Patients with Urinary Incontinence

1. Females aged ≥55 years
2. Has been living in Hong Kong for one year or more.
3. Meet the diagnostic criteria for SUI, UUI, or MUI, and the symptoms of urinary incontinence have persisted for at least 6 months.
4. Able to understand and follow written and verbal instructions in Chinese or English.
5. Provide informed consent voluntarily after being fully informed

6. Exclusion Criteria for Patients with Urinary Incontinence

1. Diagnosed with types of urinary incontinence other than stress, urge, or mixed urinary incontinence, including those secondary to neurological or systemic diseases (such as post-stroke, post-spinal cord injury, multiple sclerosis, Alzheimer's disease, Parkinson's disease, or uncontrolled diabetic peripheral neuropathy), as well as the overflow incontinence.
2. Active or structural urogenital diseases (such as unrepaired vesicoureteral reflux, congenital urethral malformations, urogenital fistula, urethral diverticulum, or active pelvic malignancies).
3. Deemed by researchers to be unable to cooperate with assessments due to severe mental or physical illness.

7. Eligible Urinary Incontinence Patients for Bio-Sample Collection

1. The first 300 urinary incontinence patients (100 each with SUI, UUI, and MUI) enrolled in the study.
2. No chronic comorbidities (except for well-controlled hypertension, defined as systolic blood pressure below 140 mmHg and diastolic blood pressure below 90 mmHg, and hyperlipidemia), including neurological disorders (central nervous system injury, motor neuron diseases, neurodegenerative diseases), diabetes, connective tissue diseases, psychiatric disorders, severe cardiovascular or cerebrovascular diseases, and severe liver or kidney diseases.
3. Not using medications that affect urination or gut microbiota (including but not limited to thiazolidinediones, sodium-glucose cotransporter-2 inhibitors, anticholinergics, α- and β-adrenergic blockers, α- and β-adrenergic agonists, diuretic antihypertensives, antihistamines, muscarinic receptor antagonists, calcium channel blockers, angiotensin-converting enzyme inhibitors, hormone medications, neurotransmitter-related drugs, gut microbiota modulators, etc.).

8. Inclusion Criteria for Healthy Volunteers

1. Female, aged ≥55 years;
2. Has been living in Hong Kong for one year or more;
3. Able to understand and follow written and verbal instructions in Chinese or English;
4. Fully informed and voluntarily signs the informed consent form.

9. Exclusion Criteria for Healthy Volunteers

1. Meet the diagnostic criteria for urinary incontinence;
2. Has a history of involuntary urine leakage, or has sought medical consultation for symptoms related to urinary incontinence;
3. Has chronic comorbidities (except for well-controlled hypertension, defined as systolic blood pressure below 140 mmHg and diastolic blood pressure below 90 mmHg, and hyperlipidemia).
4. Uses medications that affect urination or gut microbiota (including but not limited to thiazolidinediones, sodium-glucose cotransporter-2 inhibitors, anticholinergics, α- and β-adrenergic blockers, α- and β-adrenergic agonists, diuretic antihypertensives, antihistamines, muscarinic receptor antagonists, calcium channel blockers, angiotensin-converting enzyme inhibitors, hormone medications, neurotransmitter-related drugs, and gut microbiota modulators, etc.).
5. Deemed by researchers to be unable to cooperate with assessments due to severe mental or physical illness.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urinary incontinence group: Aged ≥55 years; Has been living in Hong Kong for one year or more; Meet the diagnostic criteria for MUI, UUI, or MUI defined by the International Continence Society (ICS); Able to understand and use Chinese or English; Signed the informed consent form.
  Healthy group: Aged ≥55 years; Has been living in Hong Kong for one year or more; Never went through urinary incontinence and never consult the doctor for suspect urinary incontinence related symptoms; No chronic comorbidity (expect for well-controlled hypertension and hyperlipidemia); Not taking medications that affect urination or gut microbiota; Able to understand and use Chinese or English; Signed the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of each urinary incontinence (UI) subtype (SUI, UUI, MUI) among older women with UI in Hong Kong | Baseline visit and 1-week diaries
  Percentage of participants diagnosed with SUI, UUI, or MUI, determined by standardized clinical assessment (1-hour pad test, bladder diary, ICS/EAU criteria).
Distribution of Severity among UI Patients | Baseline visit and 1-week diaries
  Proportion of UI patients classified as mild, moderate, or severe according to the Sandvik Severity Index and results of the 1-hour pad test.
Distribution of TCM Syndromes | Baseline visit
  Classification of TCM syndromes identified through standardized symptom and sign assessment, using consensus or statistical grouping approaches.
Biomarker Profiles and Their Associations with Clinical Features in UI Patients and Healthy Controls | Baseline biosample collection
  Measurement of laboratory and -omics biomarkers in blood, urine, and stool samples of UI patients (by subtype and severity) and healthy controls

SECONDARY OUTCOMES:
Urinary Incontinence Knowledge Score | Baseline assessment
  Assessment of UI knowledge using the Urinary Incontinence Questionnaire (UIQ) in patients and healthy controls.
Barriers to Incontinence Care Seeking | Baseline assessment
  Barriers to Incontinence Care Seeking Questionnaire (BICS-Q) total and subscale scores.
Quality of Life Scores (IIQ-7, ICIQ-UI-SF) | Baseline assessment
  Patient-reported impact of urinary incontinence on daily life measured with the Incontinence Impact Questionnaire-7 (IIQ-7) and International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI-SF).
Hand Grip Strength | Baseline assessment
  Hand grip strength measurement in UI patients and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Qianqian Xu, MS, RCMP, Study Director — Vincent V.C. Woo Chinese Medicine Clinical Research Institute, Hong Kong Baptist University

IPD SHARING:
Plan to Share IPD: Undecided